CLINICAL TRIAL: NCT03159013
Title: La Lambda-cyhalothrine Comme Insecticide privilégié en Milieu Agricole: étude de la toxicocinétique de Biomarqueurs Pour le Suivi de l'Exposition Des Travailleurs
Brief Title: Toxicokinetic Study of Lambda-cyhalothrin Biomarkers of Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Michèle Bouchard, Professor, Université de Montréal
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRSST-2010-0009
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Exposure to Pollution
Keywords: Pyrethroids; Lambda-cyhalothrin; Biomarkers; Toxicokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pesticide toxicokinetics- oral (Other): Exposure type: ORAL Toxicokinetics
  Interventions: Other: Exposure
- Pesticide toxicokinetics- dermal (Other): Exposure type: DERMAL Toxicokinetics
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Oral exposure: 0,025 mg/kg bw dissolved in oil, on day 1, with blood withdrawn on days 2,3,4.
  Dermal exposure: 145 µl of commercial formulation (0,25 mg/kg bw) on 40 cm2 of forearm skin for 6 hours, on day 28, with blood withdrawn on days 29,30,31.

SUMMARY:
Exposure to pyrethroid pesticides is a growing concern in the workplace especially since they are also present in the diet of the general population. It is important to monitor human exposure to these contaminants. Exposure to pyrethroids may occur by multiple routes of exposure (oral, inhalation and dermal), such that it is difficult to assess absorbed doses from external exposure assessments. Biological monitoring, which consists of measuring urinary metabolites, is now recognized by the scientific community as a preferred approach to assess exposure to this type of compound. These metabolites are biotransformation products produced in the human body from the exposure compounds. However, interpretation of these biological monitoring data requires a proper knowledge of the kinetic behavior and thus the fate of the substance of interest in the human body in order to link levels of biomarkers in individuals to actual absorbed doses. Human kinetic data are still poorly documented in the case of pyrethroids. The study in volunteers exposed to pyrethroids in controlled conditions will allow acquiring new urinary and blood profiles to refine and address uncertainties in the toxicokinetics of lambda-cyhalothrin following oral and dermal exposure. Those data will serve to build a toxicokinetic model to predict absorbed doses in workers from urinary metabolite measurements and therefore better assess health risks.

DETAILED DESCRIPTION:
Lambda-cyhalothrin is a synthetic pyrethroid pesticide widely used in Quebec to fight against pests in vegetable crops. In recent years, this pyrethroid has become one of the most used insecticides in these crops. However, there is a paucity of data on the biological behavior of this molecule in humans. Given the extensive use of this pyrethroid, it becomes essential to develop tools to properly assess exposure among workers largely in contact with pesticides during spraying or work in treated areas. Biological monitoring, which consists of measuring urinary metabolites is considered a preferred approach to evaluate absorbed doses of this type of product in the workplace, given the potentially combined exposure through the respiratory, dermal and oral routes. However, interpretation of biological monitoring data requires a good knowledge of the kinetic behavior of the substance of interest in the human body, to link biomarker levels among workers to actual absorbed doses. The overall objective of this project is to address the lack of knowledge on the toxicokinetics of biomarkers of exposure to lambda-cyhalothrin in humans for a better interpretation of routine biomonitoring data and hence health risks in exposed workers. First, a controlled kinetic study will be conducted in volunteers exposed acutely to a low oral dose of lambda-cyhalothrin (oral reference dose) followed by a cutaneous dose (of lambda-cyhalothrin formulation used by sprayers). The protocol will be similar to a previous one used by our team for toxicokinetic assessment of other pesticides. Secondly, a toxicokinetic model will be developed to simulate the kinetics of biomarkers of exposure to lambda-cyhalothrin, using data from the controlled kinetic study and based on a previous toxicokinetic model for related pyrethroids.

More specifically, volunteers will be exposed orally to 0.025 mg/kg body weight of lambda-cyhalothrin (single oral dosing). According to recent health risk assessment by the US Environmental Protection Agency (US EPA), volunteers should not incur any adverse effects relating to such dosing. Three weeks following oral dosing (to allow complete elimination of the compound from the body), the same volunteers will be exposed dermally to a lambda-cyhalothrin-based formulation used on crops. The formulation will be applied on a 40cm2 surface of the forearm at a concentration corresponding to the one used in the workplace (Matador 120EC). The treated area will not be washed for a period of 6 h. This type of application will be similar to that of exposed workers. Urinary and blood measurements of specific biomarkers of exposure to these insecticides will be performed. These biomarkers of exposure are already known from other studies and have been shown to be good bioindicators of exposure to pyrethroids. The kinetic profile will serve to link absorbed doses to blood and urinary concentrations of metabolites through time. Personal information on health status, diet and lifestyle will be documented. A total of 7 volunteers will spend a full day at the University during which they will be exposed to a low dose of pesticide. Blood and urinary samples will be collected. Four short visits of one hour will be needed for blood collections. Every urine void for a period of 84 hours will be collected in a different bottle. This whole process will be repeated twice to test two routes of exposure to this insecticide, oral (swallowed) and dermal (applied to the forearm).

The study in volunteers exposed to lambda-cyhalothrin in controlled conditions will allow acquiring new urinary and blood metabolite profiles to better understand their kinetic behavior and essential biological determinants of the observed profiles. These data can then be used in a toxicokinetic model to predict the main routes of exposure and associated absorbed doses in workers exposed to formulations containing lambda-cyhalothrin.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Caucasian origin (same group to have less genetic variability)

Exclusion Criteria:

* Pyrethroid exposure at work or home (pet, garden)
* Any kidney or liver illness

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2016-11-19 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Toxicokinetic parameters of lambda-cyhalothrin elimination after oral and dermal exposure. | 84-h post-treatment
  Elimination half-lives of biomarkers of exposure

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Bouchard, PhD, Principal Investigator — Université de Montréal; Jonathan Côté, MSc, Principal Investigator — Université de Montréal; Rania Khemiri, BSc, Principal Investigator — Université de Montréal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ratelle M, Cote J, Bouchard M. Time profiles and toxicokinetic parameters of key biomarkers of exposure to cypermethrin in orally exposed volunteers compared with previously available kinetic data following permethrin exposure. J Appl Toxicol. 2015 Dec;35(12):1586-93. doi: 10.1002/jat.3124. Epub 2015 Mar 13. PMID 25772368
- [Background] Ratelle M, Cote J, Bouchard M. Toxicokinetics of permethrin biomarkers of exposure in orally exposed volunteers. Toxicol Lett. 2015 Jan 22;232(2):369-75. doi: 10.1016/j.toxlet.2014.12.003. Epub 2014 Dec 8. PMID 25498136
- [Background] Cote J, Bonvalot Y, Carrier G, Lapointe C, Fuhr U, Tomalik-Scharte D, Wachall B, Bouchard M. A novel toxicokinetic modeling of cypermethrin and permethrin and their metabolites in humans for dose reconstruction from biomarker data. PLoS One. 2014 Feb 26;9(2):e88517. doi: 10.1371/journal.pone.0088517. eCollection 2014. PMID 24586336
- See also: U.S. EPA (2004). Lambda-cyhalothrin and an isomer Gamma-cyhalothrin; Tolerances for residues. U.S. Environmental Protection Agency. Federal Register 69(68): 18480-18489. — http://www.gpo.gov/fdsys/pkg/FR-2004-04-08/html/04-7979.htm
- See also: IRSST (2016). Développement et application d'une approche pour l'évaluation de l'exposition des travailleurs agricoles aux pyréthrinoïdes. R-936. 188 pages — https://www.irsst.qc.ca/publications-et-outils/publication/i/100895/n/evaluation-exposition-travailleurs-agricoles-pyrethrinoides